CLINICAL TRIAL: NCT03504891
Title: Cardiac MRI for Optimal Heart Failure Outcomes With CRT Upgrades
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kenneth Bilchick, MD, Associate Professor of Medicine, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRI FOR CRT UPGRADES
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Chronic Systolic Heart Failure; Paroxysmal VT

STUDY DESIGN:
Intervention Model Description: Patients will have cardiac MRI prior to CRT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MRI Prior to CRT for Upgrades (Experimental): MRI will be performed prior to CRT upgrade.
  Interventions: Diagnostic Test: MRI prior to CRT Upgrade
- MRI Prior to de novo CRT Implants (Active Comparator): MRI will be performed prior to de novo CRT implants.
  Interventions: Diagnostic Test: MRI prior to de novo CRT

INTERVENTIONS:
Diagnostic Test: MRI prior to CRT Upgrade — We will perform MRI prior to CRT to inform the optimal CRT implantation strategy in patients with existing devices undergoing upgrades versus those with de novo CRT implants. We will compare outcomes in the two groups.
  Arms: MRI Prior to CRT for Upgrades
Diagnostic Test: MRI prior to de novo CRT — We will perform MRI prior to de novo CRT implants as the comparison group.
  Arms: MRI Prior to de novo CRT Implants

SUMMARY:
This study will investigate the use of cardiac MRI in patients with standard ICDs and pacemakers to inform how cardiac resynchronization therapy (CRT) can best be implemented in these patient and which patients are the best candidates for CRT.

DETAILED DESCRIPTION:
The scientific premise of this proposal is that left and right ventricular (LV and RV) structural characteristics in patients with existing cardiac implantable electronic devices and heart failure who may benefit from an upgrade to a cardiac resynchronization therapy (CRT) device can be assessed very effectively using cardiac MRI using sequences designed for post-device imaging. Furthermore, a comparative analysis of the differences in LV/RV structural characteristics in patients with existing devices referred for CRT upgrades versus those with de novo CRT implants is expected to be very useful for developing effective strategies for optimal patient selection for CRT upgrades and implementation of CRT upgrades in appropriate patients. Patient selection for CRT upgrades is very important considering that complication rates are higher than in de novo CRT procedures and nonresponse rates are still high. With this in mind, we are performing a study of 100 patients, including 50 prospectively enrolled patients with LVEF less than or equal to 0.35 and New York Heart Association class II-III heart failure, who will be compared with an existing cohort of 50 patients with recent de novo CRT implants, pre-CRT MRIs, and response data. The 50 prospectively enrolled patients having CRT upgrades will undergo a pre-CRT cardiac MRI, pre-CRT/post-CRT echocardiography, and pre-CRT/post-CRT cardiopulmonary exercise testing. In the first aim, we will assess differences in cardiac MRI findings between CRT upgrade patients and de novo CRT patients. In the second aim, we will assess the impact of cardiac MRI findings on LV reverse remodeling and cardiopulmonary capacity in the two groups. In summary, we propose a comprehensive prospective CRT/MRI study in CRT upgrade patients with comparison to a complete MRI dataset of patients with de novo CRT implants in order to identify key differences in MRI findings in these cohorts and the impact of these MRI-based scar and activation findings on clinical outcomes. We expect that our results will have a significant public health impact for patients with heart failure referred for CRT upgrades.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing upgrade from an existing pacemaker or ICD to a CRT device.

Exclusion Criteria:

* inability to provide informed consent
* pregnancy
* presence of metal embedded in the body due to prior accident or injury, as documented by skull films or other imaging
* cerebral aneurysm clips
* cochlear implants
* other metallic implants known to be contraindications to MRI (pacemakers and ICDs are allowed)
* severe claustrophobia
* acute kidney injury
* acute renal failure
* gadolinium allergy
* abandoned leads

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
CRT Response | 6 months
  CRT Response Based on Change in LVESV After CRT

SECONDARY OUTCOMES:
Improvement in Peak Oxygen Consumption | 6 months
  Peak VO2
Improvement in Short Form (36) Health Survey | 6 months
  Assesses disability associated with heart failure. We will use the total score, which has a range of 0-100. Lower scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Bilchick, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
This research will generate MRI, echocardiographic, and cardiopulmonary exercise data in patients referred for CRT upgrades. Examples of specific data fields include the extent/distribution of myocardial scar based on late gadolinium enhancement, characterization of mechanical activation based on MRI strain imaging, baseline MRI volumetric and functional measures, changes in echocardiographic volumes and function resulting from CRT, and changes in cardiopulmonary capacity resulting from CRT.
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: Not yet available.